CLINICAL TRIAL: NCT01977274
Title: Predictive Clinical and Biological Parameters in Gynecological Cancer - GC-BIO-IPC 2013-010
Brief Title: Predictive Clinical and Biological Parameters in Gynecological Cancer
Acronym: GC-BIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GC-BIO-IPC 2013-010
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Ovarian Cancer; Endometrium Cancer; Cervix Cancer
Keywords: ovarian, endometrium, cervix cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gynecological cancer (Experimental): blood and tumor samples
  Interventions: Other: gynecological cancer

INTERVENTIONS:
Other: gynecological cancer — blood and tumor samples

SUMMARY:
Research of predictive clinical and biological factors in breast cancer : genomic, proteomic, mutation

ELIGIBILITY:
Inclusion Criteria:

* gynecological cancer suspicion
* age > 18
* signed informed consent

Exclusion Criteria:

- emergency

Exclusion criteria after histological exam Any diagnosis that is not a gynecological cancer (ovarian, cervix, endometrium).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-12; Primary Completion 2023-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
molecular alteration in gynecological cancer | average of 4 weeks after diagnosis
  gene expression level

SECONDARY OUTCOMES:
relation between molecular alteration and clinical and histological characteristics | up to 10 years
  hazard ratio between molecular alteration and clinico-histological characteristics

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli Calmettes, Marseille, France

REFERENCES:
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr